CLINICAL TRIAL: NCT07230184
Title: To Evaluate the Efficacy and Safety of Combination Therapy With B55R1 and B55R2 Compared to B55R1 Monotherapy in Patients With Non-proliferative Diabetic Retinopathy (NPDR), Focusing on Changes in Hard Exudates (HE) Over 24 Weeks.
Brief Title: To Evaluate the Efficacy and Safety of Combination Therapy With B55R1 and B55R2 Compared to B55R1 Monotherapy in Patients With NPDR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AJU Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21DR40701
Record Dates: First submitted 2025-09-22; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-Proliferative Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group(B55R1 and B55R2) (Experimental): orally twice daily
  Interventions: Drug: B55R1 and B55R2
- Control Group(B55R1 and placebo for B55R2) (Placebo Comparator): orally twice daily
  Interventions: Drug: B55R1 and placebo for B55R2

INTERVENTIONS:
Drug: B55R1 and B55R2 — After Randomization(Week 0), Participants will be administered with the drug, 2 times in a day, until end of trial(Week 24).
  Arms: Test group(B55R1 and B55R2)
Drug: B55R1 and placebo for B55R2 — After Randomization(Week 0), Participants will be administered with the drug, 2 times in a day, until end of trial(Week 24).
  Arms: Control Group(B55R1 and placebo for B55R2)

SUMMARY:
This study is planned to evaluate the efficacy and safety of combination therapy with B55R1 and B55R2 compared to B55R1 monotherapy in patients with non-proliferative diabetic retinopathy (NPDR).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 19 years or older as of the date of written consent.
2. Patients diagnosed with type 1 or type 2 diabetes.
3. Subjects with mild to severe nonproliferative diabetic retinopathy (diabetic retinopathy), grade 2-5 hard exudates
4. Subjects with a best-corrected visual acuity (BCVA) of 0.33 or higher as determined by visual acuity testing.
5. Subjects with a central retinal thickness of 350 µm or less as determined by optical coherence tomography (OCT).
6. Subjects who have received an explanation of the purpose and methods of this clinical trial and voluntarily consented to participate.

Exclusion Criteria:

1. Patients with proliferative diabetic retinopathy (diabetic retinopathy) or other causes of retinopathy.
2. Patients with uncontrolled diabetes or uncontrolled hypertension.
3. Patients with the following ocular diseases or surgical procedures:

   - Visual field defects, media opacity and ocular diseases other than diabetic retinopathywhich the investigator determines may affect the evaluation.
4. Patients who have received intravitreal and periocular steroid injections, intravitreal injection of anti-VEGF antibodies (anti-VEGF treatment), or laser photocoagulation within 12 weeks of the date of administration of the investigational drug
5. Patients taking Kallidinogenase, Vaccinium myrtillus extract, or Sulodexide
6. Patients who have experienced a cardiovascular event (unstable angina, myocardial infarction, transient ischemic attack, stroke, etc.) within 24 weeks prior to Visit 1 (participation is possible if the event occurred 24 weeks prior to Visit 1 and the patient is currently receiving medication in a stable condition)
7. Patients with severe renal impairment (renal failure requiring dialysis or (e.g., renal transplant)
8. Patients with a history of malignancy within the past 5 years from the time of screening. However, the following are eligible for clinical trial participation:

   * More than 5 years have passed since the cancer was diagnosed as cured from the screening.
   * Basal cell carcinoma, squamous cell carcinoma of the skin, thyroid cancer, or other intraepithelial neoplasms
9. Pregnant or lactating women, or those who do not agree to use adequate contraception during the clinical trial.
10. Those who have received another investigational drug within 12 weeks prior to Visit 1
11. Those who are judged by the investigator to be unsuitable for clinical trial participation due to other clinically significant medical or psychiatric findings

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects achieving a ≥1-step improvement in hard exudate grade at Week 24 | Week 24
  The proportion of subjects achieving a ≥1-step improvement in hard exudate grade at Week 24

SECONDARY OUTCOMES:
Changes in CMT as measured by OCT at Week 4, 12 and 24 | Week 4, 12 and 24
  Changes in CMT as measured by OCT at Week 4, 12 and 24
The proportion of subjects achieving a ≥1-step improvement in hard exudate grade at Week 4 and 12 | Week 4 and 12
  The proportion of subjects achieving a ≥1-step improvement in hard exudate grade at Week 4 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- AJU Pharm Co., Ltd., Seoul, South Korea